CLINICAL TRIAL: NCT03577210
Title: The Degree of Accuracy of Patient-specific PEEK Implant to Restore Chin Deficiency. Accuracy Study
Brief Title: The Degree of Accuracy of Patient-specific PEEK Implant to Restore Chin Deficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salma Hassan Abd el-Aty, Assistant lecturer, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Salma Hassan
Record Dates: First submitted 2018-05-16; First posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Chin Microgenia
Keywords: chin deficiency; chin asymmetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- computer-guided augmentation genioplasty (Other): patient-specific PEEK implant
  Interventions: Procedure: augmentation genioplasty

INTERVENTIONS:
Procedure: augmentation genioplasty — augmentation genioplasty with patient-specific PEEK implant

SUMMARY:
computer guided patient-specific PEEK implant will be used to augment patients with chin deficiency or chin asymmetry.

DETAILED DESCRIPTION:
augmentation genioplasty will be done to patients with chin deficiency or asymmetry. using cone beam CT for each patient and special soft ware "MIMICS 15" , patient-specific implant design can be done. PEEK will be milled as CAD-CAM technique to finally get patient specific PEEK implant. with patient is under General anesthesia, the implant will inserted and fixed with titanium screws. closure in two layers will be done.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patients.
* Patients with retruded chin or with chin asymmetry.
* Patients with good oral hygiene.

Exclusion Criteria:

* Patients that need skeletal procedure in the mandible, other than genioplasty, at the same time of surgery or was done within time period less than 6 months.
* Patients with medical condition that may compromise the healing process.
* Patients with medical condition that is contraindicated for general anaesthesia.
* Presence of pathological lesion related to chin area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
degree of accuracy of patient specific peek implant in chin augmentation as virtually planned using Mimics software, measuring unit (mm) mm | two weeks postoperative
  degree of accuracy of patient specific peek implant in chin augmentation as virtually planned using Mimics software, measuring unit (mm) mm

SECONDARY OUTCOMES:
patient satisfaction with postoperative chin appearance and pain: Face-Q questionnaire | 6 months postoperative
  degree of patient satisfaction using Face-Q questionnaire with score from 0-100 where 0 shows least degree of satisfaction and 100 shows best degree of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ghada abd el-monim, phd, Study Director — Cairo University
Locations (1):
- Salma Hassan, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alonso-Rodriguez E, Cebrian JL, Nieto MJ, Del Castillo JL, Hernandez-Godoy J, Burgueno M. Polyetheretherketone custom-made implants for craniofacial defects: Report of 14 cases and review of the literature. J Craniomaxillofac Surg. 2015 Sep;43(7):1232-8. doi: 10.1016/j.jcms.2015.04.028. Epub 2015 May 8. PMID 26032759
- [Background] Bertossi D, Galzignato PF, Albanese M, Botti C, Botti G, Nocini PF. Chin Microgenia: A Clinical Comparative Study. Aesthetic Plast Surg. 2015 Oct;39(5):651-8. doi: 10.1007/s00266-015-0518-4. Epub 2015 Jul 1. PMID 26130400
- [Background] Hsu SS, Gateno J, Bell RB, Hirsch DL, Markiewicz MR, Teichgraeber JF, Zhou X, Xia JJ. Accuracy of a computer-aided surgical simulation protocol for orthognathic surgery: a prospective multicenter study. J Oral Maxillofac Surg. 2013 Jan;71(1):128-42. doi: 10.1016/j.joms.2012.03.027. Epub 2012 Jun 12. PMID 22695016